CLINICAL TRIAL: NCT04596176
Title: Partnerships to Demonstrate Effectiveness of Supportive Housing for Families in the Child Welfare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chapin Hall at the University of Chicago (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Anne Farrell, Director of Research, Chapin Hall at the University of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB18-0174
Record Dates: First submitted 2020-06-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Mental Health; Physical Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Business As Usual (No Intervention): Families who were involved in the child welfare services
- Intensive Supportive Housing for Families (Active Comparator): Families who were randomly assigned in this group
  Interventions: Other: Intensive Supportive Housing Services
- Program Supportive Housing for Families (Active Comparator): Families who were randomly assigned in this group
  Interventions: Other: Program Supportive Housing Services

INTERVENTIONS:
Other: Program Supportive Housing Services — The existing statewide SH model that included routine access to housing (voucher) and case management
  Arms: Program Supportive Housing for Families
Other: Intensive Supportive Housing Services — an intensive treatment SH model with a higher dosage of case management, family teaming, and access to a vocational specialist
  Arms: Intensive Supportive Housing for Families

SUMMARY:
This was a randomized controlled trial comparing child welfare business as usual (BAU) with two levels of supportive housing (SH). To identify eligible families, a screening tool was developed that helped social workers apply a "housing lens" very early in family child welfare involvement. The study examined the extent to which implementation was faithful to the model and how well state and community partners collaborated. The research included a process evaluation, outcomes study, and economic analysis. Access to either intervention group was associated with higher family preservation and reunification, with service model intensity demonstrating minimal impact. An economic evaluation revealed that the intensive model cost the most, but the existing SH program and routine care incurred equivalent per-child costs.

DETAILED DESCRIPTION:
Supportive Housing for Families is a care management program that serves families who are experiencing child welfare needs (risk of losing custody of children or difficulty regaining custody of children) and severe housing needs. The program has been in operation for over 10 years and has been demonstrating positive outcomes for clients in terms of housing stability and family environment outcomes.

A federally funded, five-year demonstration project and evaluation focused on a new and enhanced version of the program, the Intensive Supportive Housing for Families program (ISHF). Through a three arm randomized controlled trial, this study compared clients in three groups: parents who are randomly assigned to (1) enroll in ISHF, (2) participate in the existing Supportive Housing for Families (SHF) program, and (3) receive Child Welfare Business as Usual Services. This was the first randomized evaluation of this program, and the grant required examination of whether those who participate in an enhanced version of the program, which incorporates prompt access to evidence-based interventions, vocational services, and trauma services, show superior outcomes than clients randomized to the existing program. Further, clients in both of these conditions (SHF and ISHF) were compared to those receiving child welfare services in Connecticut as usual (BAU) without a supportive housing intervention.

This research has three components: a) a process evaluation, b) a cost/economic analysis, and c) an impact analysis.

The process evaluation and cost analysis were previously completed while the project was ongoing. Now that the project has ended, the final report on all project activities has been submitted to the funder, the Administration for Children and Families.

This impact analysis addressed the following primary research questions:

1. Do clients who receive supportive housing services (SHF and ISHF interventions combined) demonstrate improved child welfare outcomes compared to those in the Child Welfare (DCF) Business as Usual (BAU) intervention?
2. Do clients who receive any supportive housing services (those in the SHF and ISHF interventions combined) demonstrate improved parental well-being compared to those in the Child Welfare (DCF) Business as Usual (BAU) intervention?
3. Do clients who receive supportive housing services (SHF and ISHF interventions combined) demonstrate improved parenting skills compared to those in the BAU intervention?
4. Do clients who receive any supportive housing services (those in the SHF and ISHF interventions combined) demonstrate increased self-sufficiency compared to those in the BAU intervention?
5. Do clients who receive any supportive housing services (those in the SHF and ISHF interventions combined) demonstrate improved child development compared to those in the Child Welfare Business as Usual intervention?
6. Do clients who receive any supportive housing services (those in the SHF and ISHF interventions combined) demonstrate improved child well-being compared to those in the Child Welfare Business as Usual intervention?

A set of secondary research questions ask: across each of these outcomes (i.e., child welfare, parental well-being, parenting skills, self-sufficiency, child development, child well-being), are there differential effects across the three intervention options, ISHF, SHF, and BAU [such that those in ISHF show greater improvement than clients in the SHF program who show greater improvement than those in BAU]?

Main outcome measures were assessed at 12, 18, and 24 months post-randomization. Housing outcomes included shelter stay and subsidy deployment. Child welfare outcomes included child removal and reunification, subsequent allegations and substantiations, and case closure.

Results: Access to either intervention group was associated with higher family preservation and reunification, with service model intensity demonstrating minimal impact. An economic evaluation revealed that the intensive model cost the most, but the existing SH program and routine care incurred equivalent per-child costs.

The PI of this research was originally at the University of Connecticut and moved to Chapin Hall. The research has concluded and the investigators are drafting a manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Families who were newly involved with the child welfare system, demonstrated high housing instability or homelessness, and evidenced high service needs.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Preservation | 2 years
  Number of children not being removed from their family
Reunification | 2 years
  Number of children being reunified with their family
Housing stability | 2 years
  Whether family remained stably housed or experienced recidivism on homelessness or near homelessness

CONTACTS AND LOCATIONS:
Overall Officials: Anne Farrell, Ph.D., Principal Investigator — Chapin Hall at the University of Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description and link to final report to the Administration on Children and Families of the Department of Health and Human Services — https://www.chapinhall.org/research/supportive-housing-ct/